CLINICAL TRIAL: NCT07119203
Title: Surgical Techniques: Robotic Versus Conventional Laparoscopic Cholecystectomy IN Benign Gallbladder Disease: A Randomized Controlled, Open, Parallel, Non-inferiority, Single-center Trial (STaRLING Trial)
Brief Title: Surgical Techniques: Robotic Versus Conventional Laparoscopic Cholecystectomy IN Benign Gallbladder Disease
Acronym: STaRLING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 333268
Record Dates: First submitted 2025-07-14; First posted 2025-08-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cholecystectomy, Robotic; Cholecystectomy, Laparoscopic; Cholecystectomy; Gallstones; Benign Gallbladder Disease
Keywords: Robotic cholecystectomy; Laparoscopic cholecystectomy; Benign gallbladder disease; Randomized controlled trial; Cost-effectiveness
MeSH Terms: conditions — Gallstones | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic cholecystectomy (Experimental): Robotic multiport cholecystectomy
  Interventions: Procedure: Robotic cholecystectomy
- Laparoscopic cholecystectomy (Active Comparator): Conventional multiport laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Robotic cholecystectomy — Robotic multiport cholecystectomy
  Arms: Robotic cholecystectomy
Procedure: Laparoscopic cholecystectomy — Conventional multiport laparoscopic cholecystectomy
  Arms: Laparoscopic cholecystectomy

SUMMARY:
This is a single-center, randomized controlled, parallel, non-inferiority trial. All adult patients with benign gallbladder disease with an indication for cholecystectomy will be assessed for eligibility and included after obtaining informed consent. A total of 276 patients will be randomized to undergo either robotic cholecystectomy (RC) or laparoscopic cholecystectomy (LC). The primary endpoint will be the incidence and severity of postoperative complications within 30 days after surgery. Secondary endpoints include perioperative outcomes, total health care utilization, health-related quality of life (HR-QoL) as assessed by patient-reported outcome measures, and cost-effectiveness. Follow-up assessments will be conducted at 7 and 30 days postoperatively.

This is the first randomized controlled trial designed to compare RC with LC in the treatment of benign gallbladder disease. The trial aims to evaluate the safety and non-inferiority of RC relative to LC, providing important evidence to guide the progress and adoption of robotic surgery in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or above 18 years;
* Benign gallbladder disease: diagnosis of gallbladder polyps or symptomatic gallstones proven on imaging (ultrasound, computed tomography (CT) scan or magnetic resonance cholangiopancreatography (MRCP));
* Capacity to give informed consent.

Exclusion Criteria:

* Minimally invasive procedure is not deemed possible by the operating surgeon;
* Evidence of acute cholecystitis;
* Known stones in the common bile duct (CBD);
* Suspicion of possible malignancy;
* Pregnancy;
* Diagnosis of liver cirrhosis (stage III or IV);
* Insufficient language skills to be able to perform the quality-of-life questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-09-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence (%) of postoperative complications within 30 days after surgery | From day of surgery up to 30 days postoperatively
  The incidence (%) of postoperative complications occurring within 30 days after surgery in patients with benign gallbladder disease. The outcome compares the total number of complications between patients treated with robotic cholecystectomy (RC) and those treated with laparoscopic cholecystectomy (LC).
Severity of postoperative complications within 30 days after surgery | From day of surgery up to 30 days postoperatively
  Complication severity will be graded using the Clavien-Dindo classification:
  1. Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.
  2. Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
     Blood transfusions and total parenteral nutrition are also included.
  3. Requiring surgical, endoscopic or radiological intervention i. intervention not under general anaesthesia ii. intervention under general anaesthesia
  4. Life-threatening complication (including central nervous system complications), requiring management in an Intensive Care Unit (ICU).
  5. Death of a patient
Frequency (%) of postoperative complications within 30 days postoperatively | From day of surgery up to 30 days postoperatively
  The frequency (%) of individual postoperative complications occurring within 30 days following surgery in patients undergoing cholecystectomy.
Comprehensive Complication Index (CCI) score within 30 days after surgery | From day of surgery up to 30 days postoperatively
  The Comprehensive Complication Index (CCI) is a validated score based on the Clavien-Dindo classification system that quantifies all postoperative complications occurring within 30 days after surgery. The score ranges from 0 (no complications) to 100 (death), reflecting the cumulative burden of morbidity per patient.

SECONDARY OUTCOMES:
Duration of the procedure (minutes) | Intraoperatively
  Two time intervals will be recorded to assess procedure duration and robotic set-up times:
  Total time spent in the operating theatre, measured as the time from patient arrival (hh:mm) to exit (hh:mm).
  Actual surgical time, measured as the time from skin incision ("knife to skin") to skin closure (hh:mm).
  Times will be recorded in minutes.
Peri-operative blood loss (millilitres) | Intraoperatively
  Peri-operative blood loss will be measured quantitatively in millilitres. Additionally, the number of tonsil swabs used during the procedure will be recorded as a qualitative indicator of blood loss.
Intra-abdominal pressure (mmHg) during surgery | Intraoperatively
  Intra-abdominal pressure will be continuously measured in millimeters of mercury (mmHg) during insufflation throughout the surgical procedure.
Incidence (%) of gallbladder perforation during surgery | Intraoperatively
  The percentage (%) of surgical procedures in which perforation of the gallbladder occurs intraoperatively.
Incidence (%) of intraoperative complications | Intraoperatively
  Percentage (%) of patients experiencing any intraoperative complication during surgery.
Technical difficulty of the procedure graded according to Nassar classification | Intraoperatively
  Technical difficulty of the procedure is graded as per Nassar et al.:
  Grade 1: Gallbladder-floppy, non-adherent; Cystic pedicle-thin and clear; Adhesions-Simple up to the neck/Hartmann's pouch Grade 2: Gallbladder-Mucocele, Packed with stones; Cystic pedicle-Fat laden; Adhesions-Simple up to the body Grade 3: Gallbladder-Deep fossa, Acute cholecystitis, Contracted, Fibrosis, Hartmann's adherent to common bile duct (CBD), Impaction; Cystic pedicle-Abnormal anatomy or cystic duct-short, dilated or obscured; Adhesions-Dense up to fundus; Involving hepatic flexure or duodenum Grade 4: Gallbladder-Completely obscured, Empyema, Gangrene, Mass; Cystic pedicle-Impossible to clarify; Adhesions-Dense, fibrosis, wrapping the gallbladder, Duodenum or hepatic flexure difficult to separate
Assessment of liver parenchyma during surgery | Intraoperatively
  Intraoperative assessment of the liver parenchyma, classified into one of the following categories based on visual and tactile evaluation by the surgeon: normal, enlarged, steatotic, or cirrhotic.
Proportion of procedures in which common bile duct (CBD) assessment was performed | Intraoperatively
  Percentage (%) of surgical procedures during which imaging-based assessment of the common bile duct (CBD) was performed. Assessment is defined as the use of on-table cholangiogram (OTC) or intraoperative ultrasound (IOUSS) for visualization of the CBD.
Proportion (%) of patients who underwent common bile duct (CBD) exploration | Intraoperatively
  Among patients in whom gallstones were identified in the common bile duct (CBD) during intraoperative assessment, the percentage (%) of cases in which CBD exploration was performed.
Use of peri-operative antibiotics | Intraoperatively
  According to current guidelines, prophylactic antibiotics are not routinely indicated. Any deviations, including type, dose, and timing of antibiotics given during surgery, will be recorded
Incidence (%) and number of drains placed during surgery | Intraoperatively
  Documentation of whether one or more surgical drains were placed intraoperatively. In cases with multiple drains, the total number of drains placed will be recorded.
Surgical perceived effort measured by Surgical Task Load Index (SURG TLX) | Intraoperatively
  Surgical perceived effort during the procedure will be assessed using the Surgical Task Load Index (SURG TLX), a surgical-specific adaptation of the NASA-TLX. The index evaluates six dimensions-mental demands, physical demands, temporal demands, task complexity, situational stress, and distractions-each rated on a 0 to 20 scale (0 = low, 20 = high). Scores will be collected from the operating surgeon immediately after the procedure.
Analgesia required in the recovery period | From arrival in recovery room until discharge from recovery
  Amount and type of analgesia administered to the patient in the post-anesthesia care unit (recovery room) from arrival until discharge from recovery. Data includes all analgesic medications given and their dosages.
Opioids prescribed upon discharge | At hospital discharge (day of discharge)
  Documentation of whether opioids were prescribed at the time of hospital discharge, including type, dose, and quantity.
Frequency (%) of same-day discharge | From surgery until discharge on the same day
  Percentage (%) of patients discharged from the hospital on the same calendar day as their surgical procedure.
Time from theatre departure to stage 3 recovery (minutes) | From theatre departure until arrival in stage 3 recovery
  Duration in minutes from the patient's departure from the operating theatre to arrival in stage 3 recovery.
Readmission rate (%) within 30 days after surgery | From day of surgery to 30 days postoperatively
  Percentage (%) of patients who are readmitted to the hospital for any cause within 30 days following surgery.
Incidence (%) of interventions needed within 30 days after cholecystectomy | From day of surgery to 30 days postoperatively
  Percentage (%) of patients requiring any additional medical or surgical interventions within 30 days following cholecystectomy.
Health-related quality of life measured by EuroQol 5D-5L (EQ-5D-5L) | At baseline (preoperative), on the day of hospital discharge, at 7 days postoperatively, and at 30 days postoperatively
  The EQ-5D-5L is a standardized patient-reported questionnaire measuring health-related quality of life. It consists of a descriptive system assessing five dimensions-mobility, self-care, usual activities, pain/discomfort, and anxiety/depression-with five severity levels each, ranging from no problems to extreme problems. Additionally, it includes a Visual Analogue Scale (EQ VAS), ranging from 0 (worst imaginable health) to 100 (best imaginable health), on which patients rate their overall health. Higher EQ-5D-5L index scores and EQ VAS scores indicate better health-related quality of life.
Gallstone-specific quality of life measured by Otago Condition-Specific Questionnaire (O-CSQ) | At baseline (preoperative) and at 30 days postoperatively
  The Otago Condition-Specific Questionnaire (O-CSQ) is a validated patient-reported questionnaire assessing gallstone-specific quality of life. It encompasses four domains: Physical Functioning (pain, dyspepsia, diet changes), Systemic Functioning (fatigue), Social Functioning (daily duties, leisure, relationships), and Emotional Functioning (mood). The O-CSQ consists of 12 items, each scored on a 5-point Likert scale (1 = no symptom burden, 5 = highest symptom burden). Higher total scores indicate a higher symptom burden and therefore poorer quality of life.
Quality of recovery measured by Quality of Recovery 15 (QoR-15) questionnaire | At hospital discharge, 7 days postoperatively, and 30 days postoperatively
  The Quality of Recovery 15 (QoR-15) questionnaire assesses postoperative recovery across five dimensions: pain, physical comfort, physical independence, emotional status, and psychological support. It consists of 15 items rated on an 11-point scale from 0 to 10. The total QoR-15 score ranges from 0 to 150, with higher scores indicating better quality of recovery.
Cost-effectiveness based on hospital costs within 30 days after surgery | From day of surgery up to 30 days postoperatively
  To assess the impact of implementing robotic cholecystectomy (RC) on hospital costs, case data will be collected and compared between the RC and laparoscopic cholecystectomy (LC) groups. This includes operative costs, admission costs, and additional treatment costs (total healthcare utilization) from the index operation up to 30 days postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication.

REFERENCES:
- [Background] Straatman J, Pucher PH, Knight BC, Carter NC, Glaysher MA, Mercer SJ, van Boxel GI. Systematic review: robot-assisted versus conventional laparoscopic multiport cholecystectomy. J Robot Surg. 2023 Oct;17(5):1967-1977. doi: 10.1007/s11701-023-01662-3. Epub 2023 Jul 13. PMID 37439902
- See also: Official trial website — https://www.starlingtrial.uk

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT07119203/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT07119203/ICF_001.pdf